CLINICAL TRIAL: NCT01276132
Title: Patient Satisfaction and Safety Outcomes After Enrollment in a Same-Day (SD) Percutaneous Coronary Intervention Program
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-291-A
Record Dates: First submitted 2011-01-10; First posted 2011-01-13 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: To Evaluate Clinical Outcomes, Safety, and Satisfaction of Patients Who Have Participated in a Same Day Outpatient Percutaneous Coronary Artery Intervention
Keywords: percutaneous coronary artery intervention; coronary disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects who are designated to receive same-day PCI
- Subjects who had been admitted to the hospital after their PCI

SUMMARY:
Subjects in this study have recently had or are scheduled for a (percutaneous coronary intervention) PCI as part of their normal, routine medical care. This procedure should restore the blood flow in the vessels of the heart.

Recent studies have shown that stable patients who undergo PCI and are discharged home after 4 hours of observation do not suffer any more complications compared to patients who stay in the hospital overnight. In addition, studies suggest that patients express increased satisfaction at being discharged after 4 hours.

The University of Chicago is one of the first US medical centers to institute a formal program of same-day discharge after PCI. This study will seek, through a analysis of medical information and satisfaction questionnaires, to assess whether this particular same-day discharge program can improve patient satisfaction and preserve patient safety.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and up
* undergoes coronary angiography in the Cardiac Catheterization Laboratory

Exclusion Criteria:

* if the subject declines participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient who presents to the Cardiac Catheterization Laboratory for coronary angiography will be given the opportunity to participate in this program. The determination on whether or not a patient is selected to undergo Same-Day PCI is based on the clinical decision of the practicing physician according to conventionally accepted inclusion and exclusion criteria. The decision on whether or not to participate in the questionnaire study will not affect any treatment decisions. The only exclusion criteria will be if the patient declines participation. The investigators would like to enroll 250 patients over a three year period.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
To evaluate clinical outcomes, safety, and satisfaction of patients who have participated in a same-day outpatient percutaneous coronary artery intervention program | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Atman Shah, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States